CLINICAL TRIAL: NCT02635035
Title: Efficacy of Lisdexamfetamine in Adults With Attention Deficit Hyperactivity Disorder (ADHD) and Sluggish Cognitive Tempo (SCT)
Brief Title: Shire SCT: Lisdexamfetamine Treatment for ADHD and SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-01288
Record Dates: First submitted 2015-11-18; First posted 2015-12-18 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lisdexamfetamine First (Experimental): In this crossover study design, participants assigned to this group will receive Lisdexamfetamine first, then placebo second
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo
- Lisdexamfetamine Second (Experimental): In this crossover study design, participants assigned to this group will receive placebo first, then Lisdexamfetamine second
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — Vyvanse (Lisdexamfetamine Dimesylate) manufactured by Shire, is a Drug Enforcement Administration (DEA) class two,sympathomimetic amine, used for the treatment of attention-deficit hyperactivity disorder. The initial adult dosage is 30mg with allowed adjustments in increments of 10mg or 20mg at weekly intervals. Subjects are initiated on these doses and then they were titrated up by 20mg with a maximum dose of 70mg.
  Other Names: Vyvanse
Drug: Placebo — Placebo looks just like Vyvanse but has no active ingredients, like a sugar pill.

SUMMARY:
The primary purpose of this study is to test the efficacy of Lisdexamfetamine in Adults With Attention Deficit Hyperactivity Disorder (ADHD) and Sluggish Cognitive Tempo (SCT). This is a placebo controlled, cross-over clinical trial of oral Lisdexamfetamine Dimesylate 30-70mg/day in adults with attention-deficit hyper-activity disorder and Sluggish Cognitive Tempo (ACT). Patients will be assigned either LDX/Placebo for 10 weeks with a two week placebo washout period.

DETAILED DESCRIPTION:
Sluggish Cognitive Tempo (SCT) describes individuals who are dreamy, spacey, slow moving, hyper active, have difficulty initiating tasks, and often seem under-motivated and under-aroused. Barkley identified nine cardinal symptoms of SCT: 1) prone to daydreaming instead of concentrating; 2) trouble staying alert/awake in boring situations; 3) being easily confused; 4) being easily bored; 5) feeling spacey/in a fog; 6) frequently feeling lethargic; 7) being under-active/having less energy than others; 8) being slow moving; 9) not processing information quickly/accurately. Individuals were identified as SCT if they had at least 5 of 9 symptoms rated often or very often on the 9-item SCT subscale from the Barkley Adult ADHD Rating Scale-IV: Self-Report (BAARS-IV; hereafter called the Barkley SCT Scale).

This is a 2 Site (NYU and Mount Sinai) Study of LDX in 50 adults with Attention Deficit Disorder (ADHD) and Sluggish Cognitive Tempo (SCT). The study will be a double-blind, 10-week, cross-over treatment trial of LDX (4 weeks; 30 - 70 mg/day) vs. placebo (4 weeks) with an intervening single- blind placebo washout period (2 weeks). During the LDX treatment period, LDX treatment will be initiated at a dose of 30mg/day at Visit 0 and can be titrated up (in the judgment of the investigator) in increments of 20mg, based upon clinical response and tolerability, to 50mg/day at Visit 1 and 70mg/day at Visit 2. Subjects receiving daily doses of 50mg or 70mg of LDX will be allowed to down titrate one dosage step of 20mg during Visits 2-4 if (in the judgment of the investigator) they are having issues in tolerability. The highest effective dose of LDX will then be maintained until Visit 4. Patients will be seen weekly throughout the trial except during placebo washout.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18-60 of all races and ethnicity.
2. Meets DSM-IV-TR criteria for a primary diagnosis of inattentive or combined type ADHD as diagnosed via the Adult ADHD Clinician Diagnostic Scale
3. For the Sluggish Cognitive Tempo+ group Must Score ≥ 5 items on the Barkley Sluggish Cognitive Tempo Scale; Must be rated 3 ("often") or ("very often") and total Sluggish Cognitive Tempo symptom score ≥ 26; must have a T-score ≥ 65 on the Metacognition Index and Motivation Subscales of the Behavior RatingInventory of Executive Function - Adult Version (BRIEF-A)
4. Impairment: must have a total score > 95th percentile on the Barkley Functional Impairment Rating Screen (Barkley Functional Impairment Scale (BFIS).
5. For the Sluggish Cognitive Tempo - group, < 5 items on the Barkley SCT Scale must be rated 3 ("often") or 4 ("very often") and total SCT symptom score < 26; must have a T-score < 65 on the Metacognition Index and Motivation Subscales of the BRIEF-A.

Exclusion Criteria:

1. Meets DSM-IV-TR criteria for a primary diagnosis of hyperactive-impulsive type ADHD.
2. Any other current psychiatric disorder, determined via the M.I.N.I , which requires pharmacotherapy treatment.
3. Current suicidal ideation or history of suicide attempts, based on the Columbia- Suicide Severity Rating Scale(C-SSRS).
4. Lifetime history of bipolar disorder or any psychotic disorder as per the M.I.N.I
5. Pregnant, breastfeeding or women planning to become pregnant.
6. Positive urine drug toxicology are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11; Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, M.D., Principal Investigator — NYU Medical College
Locations (2):
- United States (2):
  - Mount Sinai School of Medicine, New York, New York
  - New York University School of Medicine, New York, New York

REFERENCES:
- [Derived] Adler LA, Leon TL, Sardoff TM, Krone B, Faraone SV, Silverstein MJ, Newcorn JH. A Placebo-Controlled Trial of Lisdexamfetamine in the Treatment of Comorbid Sluggish Cognitive Tempo and Adult ADHD. J Clin Psychiatry. 2021 Jun 29;82(4):20m13687. doi: 10.4088/JCP.20m13687. PMID 34232582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lisdexamfetamine First | Lisdexamfetamine Second
Started | 17 | 21
Completed | 17 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine First | Lisdexamfetamine Second | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.06 (7.92) | 37.38 (11.07) | 34 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Barkley Adult ADHD Rating Scale-IV (BAARS-IV)
Description: The BAARS-IV Self-Report consists of 27 symptoms that can be rated from 1 (never or rarely) to 4 (very often). The total range of scores is 1-108; a higher score indicates ADHD symptoms at a higher frequency.
Time Frame: Baseline, 10 Weeks
Population: The intent of the study was to evaluate "the two different sequences" (that is, to compare the order of Lisdexamfetamine treatment) rather than to compare "Lisdexamfetamine" to "Placebo". Therefore, data was not collected and reported for Placebo.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lisdexamfetamine First | Lisdexamfetamine Second
Number analyzed (Participants) | 17 | 21
score on a scale | 23.27 (7.73) | 23.1 (7.4)

2. Secondary Outcome: Change in Score on Barkley Functional Impairment Scale (BFIS)
Description: BFIS is designed to evaluate possible impairment in 15 major domains of psychosocial functioning in adults. The scale for each domain is 0 to 9 where 0 represents no impairment and 9 represents highest impairment. The total range is 0-135; the higher the score, the higher the impairment.
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lisdexamfetamine First | Lisdexamfetamine Second
Number analyzed (Participants) | 17 | 21
units on a scale | 4.93 (2) | 4.88 (2.06)

ADVERSE EVENTS:
Time Frame: 11 weeks
Description: The intent of the study was to evaluate "the two different sequences" (that is, to compare the order of Lisdexamfetamine treatment) rather than to compare "Lisdexamfetamine" to "Placebo". Therefore, data was not collected and reported for Placebo.
Arm/Group | Lisdexamfetamine First | Lisdexamfetamine Second
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21
Other Adverse Events (participants affected / at risk) | 16/17 | 17/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine First (N=17) | Lisdexamfetamine Second (N=21)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 8 (13) | 5 (8)
Increased Heart Rate (Cardiac disorders) | 0 (0) | 1 (2)
Irritability (General disorders) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 0 (0) | 1 (2)
Formication (Nervous system disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (6) | 6 (8)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rapid Moving Eyes (Eye disorders) | 0 (0) | 1 (1)
Anxious/Jittery (Psychiatric disorders) | 1 (3) | 3 (4)
Heart Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Trouble Sleeping/Falling asleep (General disorders) | 3 (3) | 4 (8)
Tired (General disorders) | 1 (1) | 3 (4)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Difficulty maintaining an Erection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Change in Orgasm (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Mood Lability (Psychiatric disorders) | 0 (0) | 1 (1)
Lethargic (General disorders) | 0 (0) | 3 (3)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry Mouth (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Cold (General disorders) | 1 (2) | 1 (1)
Took Extra 50 mg Pill (Vyvanse/Placebo) (General disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Body Aches (General disorders) | 0 (0) | 1 (1)
Upper back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash on Right Hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Minor Pain in palm of Left Hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decrease Sleep (General disorders) | 1 (1) | 0 (0)
Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decreased Weight (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Sider Bite (Itchy) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
increase blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
withdrawn, subjective feelings (Psychiatric disorders) | 0 (0) | 1 (1)
over focused on work (General disorders) | 1 (1) | 1 (1)
reduced thirst (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
moody (Psychiatric disorders) | 0 (0) | 2 (2)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dry sinus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Strange Taste (General disorders) | 0 (0) | 1 (1)
itchy vagina (Reproductive system and breast disorders) | 0 (0) | 1 (1)
weird dreams (General disorders) | 0 (0) | 1 (1)
decreased creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
dry eyes (Eye disorders) | 0 (0) | 1 (1)
irritated stomach (Gastrointestinal disorders) | 1 (1) | 2 (2)
insomnia (General disorders) | 1 (1) | 4 (4)
Increased Pulse (Cardiac disorders) | 0 (0) | 1 (1)
increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
decreased memory (General disorders) | 1 (1) | 0 (0)
Sadness (Psychiatric disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0)
Mood Changes (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT02635035/Prot_SAP_000.pdf